CLINICAL TRIAL: NCT00055471
Title: A Phase IIa. Open-label, Multicenter, Dose-escalation Study to Assess the Tolerability and Pharmacokinetics of ZD4054 (Zibotentan) Given Orally Once Daily in Subjects With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 4054IL/0004
Record Dates: First submitted 2003-03-03; First posted 2003-03-04 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Prostatic Neoplasms; Metastases, Neoplasm
Keywords: prostate cancer; Metastatic prostate cancer; bone metastases
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — ZD4054

ARMS (3):
- ZD4054 10 mg (Experimental): 1 x 10 mg oral tablets once daily
  Interventions: Drug: ZD4054 10 mg
- ZD4054 15 mg (Experimental): 1 x 10 mg + 2 x 2.5 mg oral tablets once daily
  Interventions: Drug: ZD4054 15 mg
- ZD4054 22.5 mg (Experimental): 2 x 10 mg + 1 x 2.5 mg oral tablets once daily
  Interventions: Drug: ZD4054 22.5 mg

INTERVENTIONS:
Drug: ZD4054 10 mg — 1 x 10 mg oral tablets once daily
  Other Names: Zibotentan,
  Arms: ZD4054 10 mg
Drug: ZD4054 15 mg — 1 x 10 mg + 2 x 2.5 mg oral tablets once daily
  Other Names: Zibotentan
  Arms: ZD4054 15 mg
Drug: ZD4054 22.5 mg — 2 x 10 mg + 2 x 2.5 mg oral tablets once daily
  Other Names: Zibotentan
  Arms: ZD4054 22.5 mg

SUMMARY:
The primary purpose of this study is to determine the safest dose of ZD4054 (Zibotentan)in men with prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Men 18 years & older
* Confirmed diagnosis of prostate cancer with bone metastases

Exclusion Criteria:

* No more than 2 prior chemotherapy regimens
* No radiation, chemotherapy or bisphosphonates in the past 4 weeks

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2003-06; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Cleveland, Ohio
  - Research Site, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 male patients with metastatic prostate cancer and rising Prostate Specific Antigen (PSA) levels were recruited from 11th June 2003 (last subject completed on 31st October 2005). This study was conducted in 2 centres in the United States.
Pre-assignment Details: 6 of the 22 screened patients were not entered into the study as they did not fulfill the study eligibility criteria.
Groups:
- ZD4054 10 mg: ZD4054 10 mg dose: 1 x 10 mg oral tablet once daily
- ZD4054 15 mg: ZD4054 15 mg dose: 1 x 10 mg + 2 x 2.5 mg oral tablets once daily
- ZD4054 22.5 mg: ZD4054 22.5 mg dose: 2 x 10 mg + 1 x 2.5 mg oral tablets once daily
Period: Period 1: Dose Escalation Period
Arm/Group | ZD4054 10 mg | ZD4054 15 mg | ZD4054 22.5 mg
Started | 3 | 10 (Dose level given only after lower dose was successfully administered.) | 3 (Dose level given only after lower dose was successfully administered.)
Completed | 3 | 8 | 0
Not Completed | 0 | 2 | 3
Not completed — Adverse Event | 0 | 1 | 2
Not completed — Erroneously reported discont. criteria | 0 | 0 | 1
Not completed — Disease progression | 0 | 1 | 0
Period: Period 2: Extension Period
Arm/Group | ZD4054 10 mg | ZD4054 15 mg | ZD4054 22.5 mg
Started | 3 (Period 2 - attend Pts who,in the opinion of the Investigator,show benefit from treatment with ZD4054) | 6 (2 pts discontinued after completion of Period1,therefore 9 pts proceeded to participate in Period2) | 0
Completed | 3 | 6 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZD4054 10 mg | ZD4054 15 mg | ZD4054 22.5 mg | Total
Number analyzed (Participants) | 3 | 10 | 3 | 16
Age Continuous [Mean (Standard Deviation); unit: Years]
  Overall | 72.3 (3.21) | 64.6 (9.72) | 66.3 (8.08) | 66.4 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 3 | 10 | 3 | 16
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 3 | 9 | 3 | 15
  Black | 0 | 1 | 0 | 1
  Oriental | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: Centimeters (cm)] | 177.33 (4.51) | 177.10 (8.02) | 176.33 (5.03) | 177 (6.69)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 87.33 (19.035) | 107.8 (21.060) | 103.00 (35.595) | 103.06 (23.405)

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities (DLTs)
Description: DLT is defined as experiencing Common Toxicity Criteria (CTC) grade 3 or 4 headache with onset within 24 h of receiving ZD4054, CTC grade 2 rhinitis leading to the withdrawal of the subject, or other CTC grade 3 or 4 toxicity that was considered to be related to ZD4054 treatment.
  The numbers of patients with a DLT are reported.
Time Frame: Baseline to Day 29.
Measure: Number; unit: Participants
Arm/Group | ZD4054 10 mg | ZD4054 15 mg | ZD4054 22.5 mg
Number analyzed (Participants) | 3 | 10 | 3
Participants | 0 | 0 | 2

2. Secondary Outcome: Total Prostate Specific Antigen (PSA) Concentration
Description: Total Prostate Specific Antigen (PSA) concentration at Day 15 (14 doses of study treatment per patient - no dose was administered on Day 2).
Time Frame: Baseline to Day 15.
Population: All dosed patients.
Measure: Geometric Mean (Full Range); unit: ng/ml
Arm/Group | ZD4054 10 mg | ZD4054 15 mg | ZD4054 22.5 mg
Number analyzed (Participants) | 3 | 10 | 2
ng/ml | 98.454 [78.00 to 142.60] | 62.366 [6.00 to 448.90] | 56.550 [36.80 to 86.90]

3. Secondary Outcome: Change in Total Prostate Specific Antigen (PSA)
Description: Percentage change in total Prostate Specific Antigen (PSA) (ng/mL) from baseline to Day 15 (14 doses of study treatment per patient - no dose was administered on Day 2).
  Percentage change = [(measure at Day 15 - measure at baseline)/measure at baseline]*100
Time Frame: Baseline to Day 15.
Population: The analysis population includes only patients dosed with ZD4054
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | ZD4054 10 mg | ZD4054 15 mg | ZD4054 22.5 mg
Number analyzed (Participants) | 3 | 10 | 2
Percentage Change | 2.235 (15.445) | 10.986 (21.345) | 18.404 (30.132)

4. Secondary Outcome: Change in Serum Concentration of Bone Alkaline Phosphatase (ALP)
Description: Percentage change in serum concentration of Bone Alkaline Phosphatase (ALP) (ng/mL) from baseline to Day 15 (14 doses of study treatment per patient - no dose was administered on Day 2). Percentage change = [(measure at Day 15 - measure at baseline)/measure at baseline]*100
Time Frame: Baseline to Day 15.
Population: The analysis population includes only patients dosed with ZD4054
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | ZD4054 10 mg | ZD4054 15 mg | ZD4054 22.5 mg
Number analyzed (Participants) | 3 | 10 | 2
Percentage Change | -6.161 (9.616) | -9.197 (12.220) | -9.182 (10.644)

5. Secondary Outcome: Change in Serum Concentration of Procollagen Type I N Propeptide (PINP)
Description: Percentage change in serum concentration of Procollagen Type I N Propeptide (PINP) (ng/mL) from baseline to Day 15 (14 doses of study treatment per patient - no dose was administered on Day 2).
  Percentage change = [(measure at Day 15 - measure at baseline)/measure at baseline]*100
Time Frame: Baseline to Day 15.
Population: The analysis population includes only patients dosed with ZD4054
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | ZD4054 10 mg | ZD4054 15 mg | ZD4054 22.5 mg
Number analyzed (Participants) | 3 | 10 | 2
Percentage Change | 7.865 (14.625) | 20.681 (44.217) | 113.012 (51.302)

6. Secondary Outcome: Change in Serum Concentration of C-Terminal Telopeptide of Type I Collagen (CTx)
Description: Percentage change in serum concentration of C-Terminal Telopeptide of Type I Collagen (CTx) (ng/mL) from baseline to Day 15 (14 doses of study treatment per patient - no dose was administered on Day 2). Percentage change = [(measure at Day 15 - measure at baseline)/measure at baseline]*100
Time Frame: Baseline to Day 15.
Population: The analysis population includes only patients dosed with ZD4054
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | ZD4054 10 mg | ZD4054 15 mg | ZD4054 22.5 mg
Number analyzed (Participants) | 3 | 10 | 2
Percentage Change | -13.832 (19.003) | 44.855 (94.876) | 20.386 (31.094)

7. Secondary Outcome: Change in Urine Concentration of Type I Collagen-Cross Linked N Telopeptide (NTx)
Description: Percentage change in urine concentration of Type I Collagen-Cross Linked N Telopeptide (NTx) (nmol BCE/mmol Creatinine) from baseline to Day 15 (14 doses of study treatment per patient - no dose was administered on Day 2). Percentage change = [(measure at Day 15 - measure at baseline)/measure at baseline]*100
Time Frame: Baseline to Day 15.
Population: The analysis population includes only patients dosed with ZD4054
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | ZD4054 10 mg | ZD4054 15 mg | ZD4054 22.5 mg
Number analyzed (Participants) | 3 | 10 | 2
Percentage Change | -25.213 (15.389) | 2.154 (41.900) | -5.942 (34.344)

ADVERSE EVENTS:
Arm/Group | ZD4054 10 mg | ZD4054 15 mg | ZD4054 22.5 mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/10 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 10/10 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZD4054 10 mg (N=3) | ZD4054 15 mg (N=10) | ZD4054 22.5 mg (N=3)
Headache (Nervous system disorders) | 0 | 0 | 1
Intraventricular Haemorrhage (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pitting Oedema (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZD4054 10 mg (N=3) | ZD4054 15 mg (N=10) | ZD4054 22.5 mg (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Ear Discomfort (Ear and labyrinth disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Lacrimation Increased (Eye disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Tongue Discolouration (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 4 | 3
Oedema Peripheral (General disorders) | 0 | 9 | 1
Chills (General disorders) | 0 | 1 | 1
Oedema (General disorders) | 1 | 0 | 0
Face Oedema (General disorders) | 0 | 3 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0
Animal Bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthropod Sting (Injury, poisoning and procedural complications) | 0 | 0 | 1
Barotrauma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contrast Media Reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint Sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1
Weight Increased (Injury, poisoning and procedural complications) | 0 | 1 | 1
Weight Decreased (Injury, poisoning and procedural complications) | 1 | 1 | 0
Electrocardiogram Qt Corrected Interval Prolonged (Injury, poisoning and procedural complications) | 0 | 0 | 1
Haemoglobin Decreased (Injury, poisoning and procedural complications) | 0 | 0 | 1
Heart Rate Increased (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Buttock Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 9 | 3
Dizziness (Nervous system disorders) | 0 | 1 | 1
Burning Sensation (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Neuropathy (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 2 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0
Testicular Pain (Reproductive system and breast disorders) | 0 | 0 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Periorbital Oedema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
One patient received one dose of 22.5 mg and was dose reduced to 15 mg thereafter. This patient was classified into the 15 mg dose group, except for the single dose pharmacokinetic results (not posted).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days